CLINICAL TRIAL: NCT01758120
Title: A Prospective Randomized, Controlled, Open-labeled Trial of Prednisone Plus Cyclophosphamide in Patients With Advanced-stage IgA Nephropathy
Brief Title: Treatment of Prednisone Plus Cyclophosphamide in Patients With Advanced-stage IgA Nephropathy
Acronym: TOPplus-IgAN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wei Shi, clinical professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGH2012-36; GGH2012-36 (Other: GGH)
Record Dates: First submitted 2012-12-12; First posted 2013-01-01 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: IgA Nephropathy
Keywords: IgA nephropathy; Cyclophosphamide; prednisone
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Prednisone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prednisone plus cyclophosphamide (Experimental): prednisone plus cyclophosphamide: prednisone(0.5mg/kg/day*6 months) plus cyclophosphamide(1g intravenous use,per 1 month*6months)
  Interventions: Drug: prednisone plus cyclophosphamide
- prednisone alone (Experimental): prednisone alone: prednisone(0.5mg/kg/day*6 months)
  Interventions: Drug: Prednisone alone

INTERVENTIONS:
Drug: prednisone plus cyclophosphamide — 1. prednisone plus cyclophosphamide: prednisone(0.5mg/kg/day*6 months) plus cyclophosphamide(1g intravenous use,per 1 month*6months);
  2. supportive care,including ACE-I or ARBs and blood pressure control
  Arms: prednisone plus cyclophosphamide
Drug: Prednisone alone — 1. prednisone alone: prednisone(0.5mg/kg/day*6 months);
  2. supportive care,including ACE-I or ARBs and blood pressure control
  Arms: prednisone alone

SUMMARY:
Treatment of prednisone plus cyclophosphamide may be superior to treatment of prednisone alone in patients with advanced-stage IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-proven primary IgA nephropathy;
* 18-70 years old;
* elevated serum Creatinine and less than 3.0mg/dl;
* with a written consent from participants to receive prednisone and/or cyclophosphamide

Exclusion Criteria:

* diabetes;
* contraindications for the treatment of prednisone and/or cyclophosphamide;
* any treatment with steroids or immunosuppressive drugs prior to this study;
* acute deterioration of renal function(including those of glomerular origin)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
the changes of kidney function or death | 3,6 ,12, 24 and 36 months or more after treatment
  the changes of estimated glomerular filtration rate (eGFR) or a combination of reaching end-stage renal disease (ESRD) or doubling of serum Creatinine or death

SECONDARY OUTCOMES:
the changes of proteinuria | 3,6 ,12, 24 and 36 months or more after treatment

OTHER OUTCOMES:
Number of Participants with Adverse Events | 1,3,6 ,12, 24 and 36 months or more after treatment
  Number of Participants with Adverse Events; adverse events include hair loss, vomiting, diarrhea, jaundice, leukopenia, anemia, thrombocytopenia, infections, allergic reactions and hemorrhagic cystitis.

CONTACTS AND LOCATIONS:
Overall Officials: wei shi, MD PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China